CLINICAL TRIAL: NCT03081000
Title: Perioperative Hypothermia: A Multi-center Study of Incidence, Risk Factors and Preventive Measures.
Status: Completed | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: CIRB2015/2817
Record Dates: First submitted 2016-06-14; First posted 2017-03-15 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Disturbance; Temperature Regulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Aims:-

Primary:

To identify the incidence of intra-operative and post-operative hypothermia

Secondary:

To identify factors contributing to peri-operative hypothermia. To identify current anaesthetic practice in peri-operative temperature monitoring, use of active/warming measures by anaesthetists in various hospitals.

To increase awareness of the problem of IPH and guidelines available.

DETAILED DESCRIPTION:
Inadvertent peri-operative hypothermia (IPH) affects patients across all ages, occurring up to 50% in the unwarmed surgical patient. It carries significant morbidity and mortality including increased risk of myocardial infarction, bleeding, and surgical site infection, increased shivering and patient discomfort, as well as increased length of hospital stay. Guidelines have been published by the UK National Institute for Clinical Excellence (NICE) as well as the American Society of Anaesthesiologists. However, the compliance to such guidelines have been poor, and no local guidelines have been developed as yet.

A one month audit was conducted in KKH Department of Paediatric Anaesthesia in 2014 which collected data on the incidence of perioperative hypothermia in patients undergoing general anaesthesia for a variety of surgeries. This preliminary audit demonstrated a 33.7% incidence of hypothermia in PACU among 164 patients.

The investigators wish to carry out a more comprehensive audit to find out the incidence of IPH in both adult and paediatric surgical patients, identify risk factors and assess the current practice to prevent IPH across various healthcare institutions.

The study aims to find out the incidence of IPH, identify the risk factors involved and find out the current preventive measures in various local hospitals; if not already in place, bring awareness to this problem and improve patient outcomes. This is a cross-sectional observational study, aiming to recruit 4000 patients of all ages, across 5 institutions over the course of 6 months.

Patients will receive the current standard of care, as per the anaesthetist in charge, with regards to temperature monitoring, and the use of passive/active warming strategies. The method of temperature monitoring, warming or heat conservation techniques would be recorded and the patient's temperature would be measured at the recovery area post-operatively by the recovery nurse. In addition, patient demographics, surgical time, anaesthetic time, surgical procedure and method of anaesthetic, total fluids given, will also be recorded on a prospectively-designed data collection form.

ELIGIBILITY:
Inclusion Criteria:

* All cases within specified time frame under General anaesthesia (GA), Regional anaesthesia (RA), or combined General and Regional Anaesthesia (GA/RA) not involving the use of extra-corporeal circuits.

Exclusion Criteria:

* Cases done under Monitored Anaesthesia Care (MAC) or that have the use of extracorporeal circuits.

Patients that require direct admission to the intensive care unit (ICU) are also excluded as they do not transit through the recovery area.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a prospective cross-sectional observational study, aiming to recruit 4000 patients of all ages, going for surgery (day surgery/inpatient, elective/emergency). , not involving the use of extra-corporeal circuits, across 5 institutions (KKWCH, CGH, SGH, TTSH, KTPH) over the course of 6 months (oct 2015 to Mar 2016).Recruitment will be done over 1-2 months period at each site by 3 co-Investigators as they rotate through each of the anaesthetic department as part of their residency postings. A consultant site-Principal Investigator will be in charge of supervising the co-Investigators during the recruitment at each site.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Post-operative hypothermia defined as core temperature<36 degrees Celsius | Single core temperature recorded within 15 minutes upon arrival in PACU by the recovery nurse. Measurements will be taken for all recruited patients during the study period at each site.
  Mode of monitoring:
  naso/oropharyngeal/rectal temperatures for intra-opt tympanic membrane /infra-red scanner for post-opt

CONTACTS AND LOCATIONS:
Overall Officials: Shu Ying Lee, Mmed, FANZCA, Principal Investigator — KK Women's and Children's Hospital
Locations (5):
- Singapore (5):
  - Singapore General Hospital, Singapore
  - KK Women's and Children's Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Changi General Hospital, Singapore
  - Khoo Teck Phuat Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Undecided